CLINICAL TRIAL: NCT02892864
Title: Relevance of a Virtual Rehabilitation Program in Peripheral Facial Paralysis
Brief Title: Virtual Rehabilitation Program in Peripheral Facial Paralysis
Acronym: RVPF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of inclusion
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P131203; 2015-A01428-41 (Other: IDCRB)
Record Dates: First submitted 2016-07-19; First posted 2016-09-08 (Estimated); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Unilateral Peripheral Facial Paralysis
Keywords: Bell's Palsy; Peripheral facial palsy
MeSH Terms: conditions — Bell Palsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm (Active Comparator): Patients taken care in consultation within the ENT service which provides oro-myo-functional classical rehabilitation.
  Interventions: Other: Oro-myo-functional classical rehabilitation
- Experimental Virtual Arm (Experimental): Patients taken care in external consultation who receive oro-myo-functional rehabilitation through a virtual rehabilitation program targeted at the smile, in their place of living in virtual conditions.
  Interventions: Other: Neuromuscular Retraining and Virtual therapy

INTERVENTIONS:
Other: Neuromuscular Retraining and Virtual therapy — Neuromuscular retraining is a problem solving approach to treatment using selective motor training to facilitate symmetrical movement and control undesired gross motor activity (synkinesis). Treatment consists to accomplish daily massages and facial exercises. Motivation on the part of the patient is a crucial element in the success of treatment
  Arms: Experimental Virtual Arm
Other: Oro-myo-functional classical rehabilitation — Patients taken care in external consultation who receive oro-myo-functional rehabilitation through a virtual rehabilitation program targeted at the smile, in their place of living in virtual conditions.
  Patients taken care in consultation within the ENT service which provides oro-myo-functional classical rehabilitation.
  Arms: Control arm

SUMMARY:
Facial palsy can be divided into supranuclear lesion (central facial palsy) and infranuclear lesion such as Bell's Palsy, an idiopathic disease. The peripheral facial paralysis (PFP) is a frequent but little-known pathology (20 / 100 000 inhabitants in France a year). Oro-facial functions and the ability to convey emotional facial information are seriously affected by facial palsy, thereby reducing patient's quality of life. The PFP can have several repercussions on the functional, aesthetic, social, occupational and psychological levels. Evolution and prognosis depend not only on its etiology and gravity, but also on the precocity and the quality of the medical and paramedical care. It is essential to assess functional and psychological issues before beginning an adapted global therapeutic care. If these depressive symptoms can be explained by multiple factors, the inability to smile would be one of the triggering factors of depression. The facial feedback hypothesis could be one of many explications because smiling induces a positive emotional state and a feeling of well-being. In PFP, patients must cope with their difficulties to smile. Their facial behaviour affected their own emotional experiences.

The main purpose of the present study is to determine if virtual rehabilitation program is relevant compared to standard therapy. The second aim is to characterize the efficiency by analysing the time required to obtain a stable score of 4 in the Sunnybrook test. A secondary objective will be to decrease the functional and social repercussions of the facial paralysis with an intensive and targeted therapy of the smile. Furthermore, a virtual rehabilitation program will be implemented in an interactive platform.

To this end, a parallel randomized controlled trial (RCT) of the two groups will be conducted: standard therapy versus virtual rehabilitation program. RCT involves a treatment in which active participation of the patient is necessary so only the assessment will be blinded. Facial motor skills (tongue, mouth and face motricity) are measured using electronic devices, objective and subjective evaluation with pragmatic fields such as communication, emotion and quality of life. The severity of patient's facial paralysis is appraised by the House and Brackmann scale. This global assessment will be conducted before the beginning of the therapy and every 3 months during 18 months.

The patients will be recruited within the Ear, Nose, and Throat (ENT) service after a baseline assessment. Simple randomization will be used in order to establish both therapeutic groups with 45 patients in each group.

Group A: Patients taken care in consultation within the ENT service which provides oro-myo-functional classical rehabilitation.

Group B: Patients taken care in external consultation who receive oro-myo-functional rehabilitation through a virtual rehabilitation program targeted at the smile, in their place of living in virtual conditions.

The patients must have been diagnosed with unilateral peripheral facial palsy, according to House and Brackmann international classification.

Inclusion time : 18 months

Between-two-groups analysis will be conducted in order to compare a targeted and intensive implementation-intention rehabilitation such as virtual rehabilitation program to standard therapy. This virtual therapy will consist in repeating mentally movement desired, so that it will be more spontaneously executed in the every-day-life situation.

DETAILED DESCRIPTION:
Facial palsy can be divided into supranuclear lesion (central facial palsy) and infranuclear lesion such as Bell's Palsy, an idiopathic disease. The peripheral facial paralysis (PFP) is a frequent but little-known pathology (20 / 100 000 inhabitants in France a year). Oro-facial functions and the ability to convey emotional facial information are seriously affected by facial palsy, thereby reducing patient's quality of life. The PFP can have several repercussions on the functional, aesthetic, social, occupational and psychological levels. Evolution and prognosis depend not only on its etiology and gravity, but also on the precocity and the quality of the medical and paramedical care. It is essential to assess functional and psychological issues before beginning an adapted global therapeutic care. Although these depressive symptoms can be explained by multiple factors, the inability to smile would be one of the triggering factors of depression. The facial feedback hypothesis could be one of many explications because smiling induces a positive emotional state and a feeling of well-being. In PFP, patients must cope with their difficulties to smile. Their facial behaviour affected their own emotional experiences.

Time required for improvement and risk of sequelae are proportional in the severity of the paralysis (speed of installation and axonal loss). Do the patients benefiting from virtual care have a deadline of recovery faster than control patients? Does a virtual rehabilitation program, home delivered, which is targeted at the smile improve symmetric movements and reduce psychological and functional issues?

The main purpose of the present study is to determine if virtual rehabilitation program is relevant compared to standard therapy. The second aim is to characterize the efficiency by analysing the time required to obtain a stable score of 4 in the Sunnybrook test.

A secondary objective will be to decrease the functional and social repercussions of the facial paralysis with an intensive and targeted therapy of the smile. Furthermore, a virtual rehabilitation program will be implemented in an interactive platform.

To this end, a parallel randomized controlled trial (RCT) of the two groups will be conducted: standard therapy versus virtual rehabilitation program. RCT involves a treatment in which active participation of the patient is necessary so only the assessment will be blinded. Facial motor skills (tongue, mouth and face motricity) are measured using electronic devices, objective and subjective evaluation with pragmatic fields such as communication, emotion and quality of life. The severity of patient's facial paralysis is appraised by the House and Brackmann scale. This global assessment will be conducted before the beginning of the therapy and every 3 months during 18 months.

The patients will be recruited within the ENT service after a baseline assessment. Simple randomization will be used in order to establish both therapeutic groups with 45 patients in each group.

Group A: Patients taken care in consultation within the ENT service which provides oro-myo-functional classical rehabilitation.

Group B: Patients taken care in external consultation who receive oro-myo-functional rehabilitation through a virtual rehabilitation program targeted at the smile, in their place of living in virtual conditions.

Oro-myo-functional classical rehabilitation (Diels et al.):

Neuromuscular retraining is a problem solving approach to treatment using selective motor training to facilitate symmetrical movement and control undesired gross motor activity (synkinesis). Treatment consists to accomplish daily massages and facial exercises (ten minutes per day). Motivation on the part of the patient is a crucial element in the success of treatment Tools such as feedback and specific mirror exercises provide augmented sensory information to enhance neural adaptation and learning. Patient education is the most basic aspect of the therapeutic process. The facial therapist provides training in basic facial anatomy, physiology and kinesiology pertinent to each patient's specific situation.

Treatment is based on functional profile. Techniques will be used to facilitate movement and inhibit abnormal patterns refine motor control, coordination and complexity of movement. The specific objectives of the reeducation are to mobilize the paralyzed hemiface and to avoid the over-investment of the healthy hemiface via the relaxation. Focus: to inhibit the abnormal over-activity rather than to strengthen muscles. Although each patient's program differs, there are common aspects in the treatment of all patients.

The technique is based on three fundamental principles:

* Slow execution to maintain inhibition as exercise increases - minimal, incremental movements. Initiating movements slowly and gradually allows the patient to observe and modify the angle, strength and speed of the excursion as it occurs. As a result, new motor control strategies are systematically developed and learned.
* Small movements enough to mimic expressive movements and decrease overflow. Small movements preserve isolated responses of the facial muscles by limiting motor unit recruitment to those muscles targeted.
* Symmetry. Patients are instructed in symmetrical exercise of movements to reinforce the normal physiological response.

Clinic treatment sessions are designed to identify, develop and refine the movement patterns that will be of greatest benefit to each patient. Patients practice these movement patterns repeated in the clinic to assure accuracy. Through the home program, patients consistently practice the strategies learned in the clinic.

Virtual Rehabilitation program:

It's in the e-health context that virtual rehabilitation program should be considered. E-health is a recent term for healthcare practice supported by electronic processes and communication. E-health is becoming more and more as the solution for universal access to high quality care.

The virtual rehabilitation program is a computerized rehabilitation, remotely managed by the therapist. This rehabilitation would meet patients' and therapists' expectations with the aim of dealing with the lack of therapists trained in the specific rehabilitation of the PFP. It will avoid too frequent and binding travels of the patients. Indeed, kilometric average of paralyzed patients taken care in the ENT service in Pitié-Salpêtrière is about 88 km. This virtual rehabilitation program would then meet the requirements of the law '' Hospital, Patient, Health and Territory '' of July 29th, 2009.

This virtual rehabilitation could also help patients to stay motivated by involving them actively in the rehabilitation process. In fact, the patient is an autonomous actor of his own rehabilitation. Furthermore, visual feedback provided by the avatar will help them to execute movements in a proper way

Patient data is transferred to the therapists. At distance, the clinician is able to straighten the exercises to execute and to update the method while waiting for the next patient consultation.

The patient will be in front of his screen and the avatar will produce '' praxies'' according to the evolution and the severity of the PFP (House and Brackmann scale). It is recommended to observe the avatar repeatedly (three times a day for two weeks) so that, the patient will learn the appropriate motor schemes. Then, the patient will apply the '' implementation-intention '' technique in order to find the movement in any circumstances. This technique consists in repeating mentally in advance the deliberate movement, so that it will be executed more spontaneously in every-day-life situation.

Administration tool presents two sectors: it allows on one hand to consult the recorded patients (addition, modifications, consultation of the exercises video, rehabilitation management and updating, indication of the next recommended exercises, addition of a note for the next session...). On the other hand, it allows to manage the exercises which include a number of poses. For every pose, maintaining poses time and number of iterations of the pose is indicated.

Digital, still sub-used technology, represents a real potential to improve professional practices.

The patient training tool is a Windows run-time software which connects to the database and downloads the exercises of the session. This connexion involves an automatic identification. The software begins with a message posted by the therapist. Then, a simple interface, including a half-screen posting what sees the webcam and another half-screen showing the avatar which serves as a model for the training sessions. The patients are able to record their own pose and to try again if they need to. In the end, a message indicates the end of the current session.

Statistical Analysis:

Between-two-groups analysis will be conducted in order to compare a targeted and intensive implementation-intention rehabilitation such as virtual rehabilitation program to standard therapy. This virtual therapy will consist in repeating mentally movement desired, so that it will be more spontaneously executed in the every-day-life situation.

All the quantitative variables, as the Sunnybrook score, the bilabial strength, the House-Brackmann score, the MADRS score and the Quality of Life score will be described by their average score, standard deviation, median score, minimum and maximum score. Category-specific variables as Spielberg stress scale, Mouth-tongue-face motricity assessment will be described by their frequencies and their percentages. Missing data will be taken into account in these calculations Reliable intervals in 95% will be supplied when it will be necessary.

Percentages in both groups will be compared by Pearson X2 tests or Fisher tests according to the distribution. Continuous data will be compared by Student tests or Mann-Whitney tests, according to their distribution. P-values must be lower than 0,05 in order to be considered as statistically significant..

Analyses will be realized in intention to treat, under the responsibility of the Biostatistics pole of Clinical Research Unit (URC) Pitié-Salpêtrière Charles Foix, with the software SAS 9.2 (SAS(AIRLOCK,SIEVE,AIRLOCKS) INSTITUTE, CARY, NC).

ELIGIBILITY:
Inclusion Criteria:

* Man or women ≥ 18 years
* Diagnosed with UNILATERAL peripheral facial palsy according to the criteria of the International Classification of House and Brackmann (HB) between grades III and VI.
* Informed and having signed the consent form
* Patient who has a computer with webcam and an internet connection
* Affiliated to social security scheme (not accepted AME)

Exclusion Criteria:

* Major unable, protected, deprived of freedom
* Patients with facial palsy with a tumoral origin
* Patients with uncorrected vision problems
* Patient who have had botulinum toxin injections .
* Patient who have underwent rehabilitation of type electrical stimulations
* Patient who has a facial diplegia , a graft of the face or a grade I or II House and Brackmann (HB) .
* Patient who underwent rehabilitation of the paralyzed face

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-10-24 (Actual); Primary Completion 2018-02-20 (Actual); Study Completion 2018-03-07 (Actual)

PRIMARY OUTCOMES:
Facial muscle function using Sunnybrook Facial Grading System (SFGS). | 18 months
  Assessment of facial muscle function using SFGS was performed blindly by a therapist who was unaware of the type of rehabilitation program which the patient had received (virtual or standard therapy). The time required to obtain a stable score of 4 under the SFGS will be compared between both therapies.

SECONDARY OUTCOMES:
Functional and psychological impacts using a specific questionnaire | 18 months
  Assessment of the functional and psychological impacts of the facial paralysis by using a specific quality-of-life questionnaire graduated from 0 to 3 per item and up to 99 points maximum score.
Implementation of a virtual rehabilitation platform using questionnaires | 18 months
  The relevance of a virtual rehabilitation will be assessed by specific questionnaires. Moreover, time-comparison to obtain a stable score of 4 at the Sunnybrook Grading Scale will be conducted between both therapies.

CONTACTS AND LOCATIONS:
Overall Officials: Georges LAMAS, PUPH, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- APHP - Pitié-Salpêtrière Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Diels HJ, Combs D. Neuromuscular retraining for facial paralysis. Otolaryngol Clin North Am. 1997 Oct;30(5):727-43. PMID 9295250